CLINICAL TRIAL: NCT00425659
Title: Evaluation of New Diagnostic and Treatment Algorithm for Obstructive Sleep Apnea in High Risk Population in Hong Kong
Brief Title: Evaluation of New Diagnostic and Treatment Algorithm for Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Doctor, CUHK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CRE-2006.404-T
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Sleep Apnea
Keywords: Health utility; Home sleep study
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3 (Active Comparator)
  Interventions: Device: home CPAP titration (Autoset)
- 1 (Experimental)
  Interventions: Device: home sleep study
- 2 (Other): usual practice
  Interventions: Device: CPAP

INTERVENTIONS:
Device: home sleep study — different in algorithm arrangement for diagnosing sleep apnea
  Other Names: different algorithm arrangement
  Arms: 1
Device: home CPAP titration (Autoset) — continuous positive airway pressure device for treatment of sleep apnea
  Other Names: Autoset
  Arms: 3
Device: CPAP — usual practice
  Arms: 2

SUMMARY:
Newer home sleep study device and algorithm provides an alternative for inpatient sleep study and improve the service provides to patients

DETAILED DESCRIPTION:
Purpose: Assess different potential algorithms to improve the service and cost utility for diagnosis and treatment of obstructive sleep apnea syndrome (OSAS) in patients with high pretest probability in Hong Kong.

Hypothesis: Newer home sleep study device and algorithm provides an alternative for inpatient sleep study Design: Prospective randomized study Subject: High pretest probability of OSAS patients referred to a tertiary centre.

Study instruments: a portable sleep study device, AutoCPAP and inpatient sleep monitoring system.

Interventions: comparison between 3 different algorithms of health service for OSA patients would be made: conventional in-patient sleep study, empirical treatment and home sleep study.

Main outcome measures: The primary outcome is the validity of the home sleep study device compare to inpatient sleep study. The secondary outcomes are the relative efficacy of different algorithms and the numbers of failed procedures in each algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with high pretest probability of OSAS, i.e. ESS > 10 or symptomatic patients, with BMI > 23 and/or cranial facial features associated with OSA, as assessed by the attending respiratory physician in the respiratory clinic.
* Patients aged between 18-65 years who agree to participate in the study.

Exclusion Criteria:

* Pregnant women
* Patients who refuse signing consent of the study
* Do not have high pretest probability of OSAS
* Refuse to have home sleep study
* Refuse any treatment offered; or
* Could not comply with the set up of home study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Validity of the new home sleep study device compare with conventional inpatient sleep study | 1 year

SECONDARY OUTCOMES:
The relative efficacy between different algorithm | 1 year
Failure rates in different algorithms which need to switch to the conventional algorithm | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kin W To, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, China